CLINICAL TRIAL: NCT02043431
Title: Genetic and Electronic Medical Records to Predict Outcomes in Heart Failure Patients
Brief Title: Electronic Medical Records and Genomics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Other Study IDs: EMR-01
Record Dates: First submitted 2014-01-20; First posted 2014-01-23 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-01

CONDITIONS: Heart Failure
Keywords: Heart failure; Electronic medical records; Genomics; Biobank
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Whole blood, urine. Exhaled acethone.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to develop a biobank containing samples of 2,000 patients treated in a tertiary cardiology hospital containing electronic medical records and genetic data in genome-wide scale for performing genetic association studies for validation and development of medical decision routines that help the clinical management of heart failure patients.

DETAILED DESCRIPTION:
Patients between 18 and 80 years old with heart failure diagnosis of different etiologies and left ventricular ejection fraction < 50% in the past 2 years will be eligible for enrollment on the cohort. After consent, patients will be submitted to clinical baseline, echocardiographic, cardiography impedance and biochemical evaluation. Study data will be collected and managed using Research Electronic Data Capture (REDCap) tools. The follow up will take place every 6 months to assess cardiovascular outcomes (all-cause mortality, cardiovascular mortality, hospitalization for worsening heart failure and current medication use). Initial analytical strategy will focus on the establishment of the accuracy of electronic medical records extraction protocols for main predictor factors of morbidity and mortality in heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years old
* Heart failure diagnosis of different etiologies
* Left ventricular ejection fraction < 50% in the past 2 years

Exclusion Criteria:

* Patients with impaired cognition due to advanced dementia syndrome or severe psychiatric disorder
* Patients without telephone access
* Patients that refused to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The elegible individuals are patients of a tertiary cardiology hospital
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-08; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | six and twelve months after inclusion.
  Deaths for all causes after 6 months of inclusion. Deaths for all causes after 12 months of inclusion

SECONDARY OUTCOMES:
cardiovascular mortality | six and twelve months after inclusion.
  Deaths for cardiovascular cause after 6 months of inclusion. Deaths for cardiovascular cause after 12 months of inclusion.

OTHER OUTCOMES:
Hospitalization for any cause | six and twelve months after inclusion.
  necessity of hospital care in 6 and 12 months of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre C Pereira, MD, PhD, Principal Investigator — Heart Institute - Clinical Hospital - University of São Paulo Medical School
Locations (1):
- Heart Institute - Clinical Hospital - University of São Paulo Medical School, São Paulo, Brazil